CLINICAL TRIAL: NCT07030530
Title: The Effect of Virtual Reality Video and Mandala Coloring Activity on Anxiety Levels, Satisfaction and Non-Stress Test Results of Pregnant Women
Brief Title: Virtual Reality Video and Mandala Coloring Activity on Anxiety Levels, Satisfaction and Non-Stress Test Results of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Keskin Töre (Other)
Responsible Party: Sponsor-Investigator, Fatma Keskin Töre, Assistant Professor, PhD, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/17
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; State Anxiety
Keywords: State Anxiety; Pregnancy; Mandala Coloring; Non-Stress Test; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Glasses Group (Experimental): Virtual Glasses Group; Pregnant women in the virtual reality group will be shown a virtual reality video in VR mode via smartphone during the NST procedure (with the pregnant woman lying on her left side). It will be watched with virtual reality glasses containing nature sounds (streams, birds, etc.). Pregnant women will be informed about the use of virtual reality goggles before being shown the virtual reality video and will be asked to stop watching the video if they feel any discomfort. Virtual reality videos are recommended to be watched for 5-20 minutes as they may cause nausea and vomiting. Since this study includes pregnant women, it is planned to play the virtual reality videos for 5-10 minutes.
  Interventions: Device: Virtual Glasses Group
- Mandala Coloring activity group (Experimental): Mandala Coloring activity group; In studies examining the effect of art therapy on the reduction of psychological symptoms, it has been shown that the use of round patterns is more effective in symptom management.(24) In line with these studies, ready-made mandala coloring templates with round shapes will be used in our study (25,26). Each participant will be asked to choose one of the mandala coloring templates. Each participant will be given colored pencils and asked to color the mandala template of their choice during the NST (27,28).
  After the procedure is completed, the pregnant women will be asked the State Anxiety Scale, VAS-Satisfaction form and the NST Findings Record Form will be completed by the researcher.
  Interventions: Other: Mandala Coloring activity group;
- Control Group (No Intervention): Pregnant women in the control group will undergo standard outpatient clinic practice. Pregnant women in the control group will be asked Personal Information Form and State Anxiety Scale form questions in the pretest. After the procedure is completed, the pregnant women will be asked the State Anxiety Scale, VAS-Satisfaction form in the post-test and the NST Findings Record Form will be completed by the researcher.

INTERVENTIONS:
Device: Virtual Glasses Group — Virtual Glasses Group; Pregnant women in the virtual reality group will be shown a virtual reality video in VR mode via smartphone during the NST procedure (with the pregnant woman lying on her left side). It will be watched with virtual reality glasses containing nature sounds (streams, birds, etc.). Pregnant women will be informed about the use of virtual reality goggles before being shown the virtual reality video and will be asked to stop watching the video if they feel any discomfort. It is recommended to watch virtual reality videos for 5-20 minutes because they may cause nausea and vomiting (23). Since this study includes pregnant women, it is planned to play the virtual reality videos for 5-10 minutes.
  Arms: Virtual Glasses Group
Other: Mandala Coloring activity group; — Mandala Coloring activity group; In studies examining the effect of art therapy on the reduction of psychological symptoms, it has been shown that the use of round patterns is more effective in symptom management. In line with these studies, ready-made mandala coloring templates with round shapes will be used in our study. Each participant will be asked to choose one of the mandala coloring templates. Each participant will be given colored pencils and asked to color the mandala template of their choice during the NST
  Arms: Mandala Coloring activity group

SUMMARY:
Non-stress testing (NST) is one of the most commonly used non-invasive tests to assess fetal health. NST is widely used because it is non-invasive and easy to interpret. However, although it is a painless procedure, pregnant women may experience anxiety during the procedure. The high level of anxiety experienced by the pregnant woman during the NST procedure affects the test result and may increase the rate of non-reactive NST, leading to misinterpretation. These false positive rates of NST lead to an increase in cesarean section rates. Recent studies have shown that methods that increase fetal movements and shorten the duration of NST are used. When the literature is examined, it is seen that non-pharmacological methods such as music therapy, virtual reality and abdominal touching applied during the NST procedure reduce the anxiety of pregnant women and positively affect the NST results. With this proposed project, it is aimed to determine the Effect of Virtual Reality Video and Mandala Coloring Activity on Anxiety Levels, Satisfaction and Non-Stress Test Results of Pregnant Women.

The study is a randomized controlled experimental type study in pretest-posttest design and the population of the study will consist of pregnant women who applied to Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital Obstetrics and Gynecology Outpatient Clinic and were referred to NST. Simple randomization method will be used while sampling the pregnant women. The power analysis was performed under 95% power (1-β), number of groups=3 and α=0.05, and in the light of these parameters, it was concluded that a sample size of at least 90 participants was required for this study. In case of data loss, it was envisaged to increase the sample size by 20%. Accordingly, the project was planned to be conducted with a total of n=108 participants, with 36 pregnant women in each group. After the ethics committee permission, institutional permission will be obtained from Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital. Data will be collected using the "Personal Introduction Form", "State Anxiety Scale", "NST findings record form" in which NST findings are recorded, and Visual Analog Scale-Satisfaction Form to evaluate their satisfaction after NST.

DETAILED DESCRIPTION:
In the first part of the study, pregnant women who apply to Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital Obstetrics and Gynecology Outpatient Clinic and are referred to NST and meet the inclusion criteria will be informed about the project and verbal and written consent will be obtained. In this direction, survey questions will be directed to pregnant women who agree to participate in the study. In the study, pre-test data will be obtained with 13-question Participant Introduction Form and 20-question State Anxiety Scale forms. Post-test data will be obtained after the NST procedure is completed for the experimental groups, the researcher will ask the State Anxiety Scale, VAS-Satisfaction form by face-to-face interview method and the NST Findings Record Form will be filled by the researcher.

and the explanations made to the pregnant women before the procedure will be made in a room outside the NST room.

Randomization Pregnant women included in the study will be randomized with the single-blinded randomized rule. Randomization will be done by using the random integer generator method in the numbers subheading of the random.org website, and three-group columns will be created with numbers from 1 to 108. At the beginning of the study, lots will be drawn to determine which of the 3 columns will be the experimental groups and which will be the control group. When there is a participant who meets the inclusion criteria, the participant will be included in whichever group the next number is in.

Data Collection Tools Data will be collected using the Personal Introduction Form, which determines the socio-demographic and obstetric characteristics of women and their knowledge about NST, the State Anxiety Scale, the NST Findings Record Form, which includes the findings related to NST, which allows the researchers to evaluate the NST result of pregnant women, and the Visual Analog Scale (VAS) - Satisfaction Form to evaluate their satisfaction after NST.

Personal Introduction Form This form was created by the researchers to determine women's sociodemographic (age, educational status, etc.), obstetric characteristics (pregnancy, abortion and number of living children) and knowledge about NST (receiving information about NST before, from whom they received the information, reason for NST withdrawal, etc.).

State Anxiety Scale (SAS) The adaptation of the State-Trait Anxiety Scale, which was developed by Spielberg et al. in 1970 to measure anxiety level, into Turkish was performed by Öner and Le Compte (1983). The scale consists of two parts and the State Anxiety part was used in this study. There are 20 statements in the scale . The scales include both direct statements and inverted statements. While direct statements express negative emotions, inverted statements reflect positive emotions. In the State Anxiety Scale, these reversed statements are items numbered 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The statements in the scale are answered by marking (1) not at all, (2) a little, (3) a lot, and (4) completely in order to evaluate emotions or behaviors according to the severity of the experiences. The total score obtained varies between 20 and 80. A high score on the scale indicates a high level of anxiety. The Cronbach alpha value of the scale was found between 0.94 and 0.96 .

NST Findings Record Form The NST Findings Record Form is a form used by researchers to evaluate the NST results of pregnant women. This form contains data in which the findings of NST of pregnant women are recorded .

Evaluation of the NST Findings Record Form; NST results of pregnant women were evaluated by the researchers. As reactive NST, the result of the test will be accepted as reactive NST in the presence of at least two accelerations lasting at least 15 seconds and 15 beats/minute more than the baseline beat within 20 minutes of electronic fetal heart rate tracings . As nonreactive NST, the result of the test will be considered as nonreactive NST in the absence of at least two accelerations lasting at least 15 seconds and lasting more than 15 beats/min more than the baseline beat within 20 minutes of printing electronic fetal heart rate tracings, in the presence of severe variable deselerations and late deselerations, or in the development of continuous fetal tachycardia of 160 beats/min or more when the baseline tracings are normal .

Visual Analog Scale (VAS)- Satisfaction Form The scale developed by Price et al. (1983) is a very simple, easy-to-administer measurement method used to measure subjective experiences. It is a measurement tool that is evaluated by individuals marking a horizontal or vertical line of 10 cm or 100 mm, with one end indicating "very good" and the other end indicating "very bad". This line is only straight

ELIGIBILITY:
Inclusion Criteria:

To be over 18 years of age,

* Not having any chronic or metabolic disease (completely healthy pregnant women)
* Not having any psychiatric illne

Exclusion Criteria:

* -Multiple pregnancy
* Contraction on NST communication and visual impairment, uterine contraction as a result of NST,
* Have any chronic disease (such as diabetes mellitus, hypertension, heart failure),
* Have pregnancy complications (such as pre-eclampsia, gestational diabetes, Rh incompatibility),
* History of infertility and conceived with assisted reproductive techniques,
* The fetus has an identified problem (such as anomaly, intrauterine growth retardation and cardiovascular disease),
* Pregnant women who provided false or incomplete information were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The Effect of Virtual Reality Video and Mandala Coloring Activity on Non-Stress Test Results | 20 minutes later
  Reactive Non-Stress Test Results

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam Üniversitesi, Kahramanmaraş, Turkey (Türkiye)